CLINICAL TRIAL: NCT04020718
Title: Engagement With an Adaptive Mobile Health Smoking Cessation Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gina Kruse, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019A005710
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Tobacco Use Cessation
Keywords: mobile health
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: Pilot sequential multiple assignment randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early assessment (Experimental): Patients are assessed for response to brief telephone advice plus a tailored text message program at 4 weeks post-randomization. Response is based on self-reported 7-day point prevalence abstinence. Non-responders are randomized to 4 weeks of mailed nicotine patches and/or lozenges (NRT) or 4 weeks of mailed NRT plus proactive telephone coaching.
  Interventions: Behavioral: Brief telephone advice plus tailored text messages; Drug: Mailed nicotine replacement therapy; Behavioral: Proactive telephone coaching
- Late assessment (Experimental): Patients are assessed for response to brief telephone advice plus a tailored text message program at 8 weeks post-randomization. Response is based on self-reported 7-day point prevalence abstinence. Non-responders are randomized to 4 weeks of mailed nicotine patches and/or lozenges (NRT) or 4 weeks of mailed NRT plus proactive telephone coaching.
  Interventions: Behavioral: Brief telephone advice plus tailored text messages; Drug: Mailed nicotine replacement therapy; Behavioral: Proactive telephone coaching

INTERVENTIONS:
Behavioral: Brief telephone advice plus tailored text messages — All patients are offered brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training and a text message program tailored to readiness to quit and quit date. Content is personalized with user's name and Massachusetts General Hospital resources.
Drug: Mailed nicotine replacement therapy — Patients who report continued smoking at Early or Late assessment (depending on random assignment) will be offered a 4 week supply of patches and/or lozenges dosed according to package instructions (patches dosed according to cigarettes smoked per day and lozenges dosed according to time to first cigarette).
Behavioral: Proactive telephone coaching — Patients who report continued smoking at Early (4-week) or Late (8-week) assessment of response will be randomized to receive proactive telephone coaching or not. Proactive coaching will consist of an attempt to reach the patient by telephone in order to review quit activities, provide information about locally available pharmacologic and behavioral treatment options and information sharing with patient's primary care provider. The coach is trained in core Tobacco Treatment Specialist activities.

SUMMARY:
This is a pilot sequential multiple assignment trial (SMART) to understand the optimal timing to assess response to our smoking cessation text message intervention and to measure how adding medications alone compares to adding medications and telephone coaching for those who continue to smoke. This study aims to assess the feasibility of a SMART of a proactively offered text message intervention for smokers in primary care that compares early (4 weeks) versus late (8 weeks) assessment of treatment response and the addition of nicotine replacement therapy (NRT) alone or with telephone coaching for non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Smoking status of current smoker in structured field of electronic health record (EHR)
* Language listed as English in EHR
* Massachusetts General Hospital patient, Partners healthcare primary care provider (PCP)
* PCP visit in the past 2 years
* Mobile telephone number listed in EHR

Exclusion Criteria:

* Not a current daily smoker defined as not having smoked ≥100 cigarettes in lifetime or self-report of less than daily current smoking
* Pregnant, planning to become pregnant in the next 3 months, or breastfeeding.
* Past 30-day use of nicotine replacement therapy, bupropion, or varenicline.
* Past 30-day use of Massachusetts state quit-line or SmokefreeTXT programs
* Prior serious adverse reaction to the nicotine patch or lozenge defined as any reaction that was life-threatening, required hospitalization, or other clinical evaluation
* Ever had an allergy to nicotine patch
* Weight < 100 pounds
* Unstable coronary disease
* Unstable arrhythmia
* Dementia or active psychosis or schizoaffective disorder
* Willing and able to receive and participate with a text message program for up to 12 weeks
* Unable to read English or unable to write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina R Kruse, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massacusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kruse GR, Joyce A, Yu L, Park ER, Neil J, Chang Y, Rigotti NA. A pilot adaptive trial of text messages, mailed nicotine replacement therapy, and telephone coaching among primary care patients who smoke. J Subst Use Addict Treat. 2023 Feb;145:208930. doi: 10.1016/j.josat.2022.208930. Epub 2023 Jan 6. PMID 36880910

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Assessment: Participants are assessed for response to brief telephone advice plus a tailored text message program at 4 weeks post-randomization. Response is based on self-reported 7-day point prevalence abstinence. Those who continue to smoke are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of mailed NRT plus proactive telephone coaching.
  Brief telephone advice plus tailored text messages: All patients are offered brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training and a text message program tailored to readiness to quit.
  Mailed nicotine replacement therapy: Patients who report continued smoking at Early or Late assessment (depending on random assignment) will be offered a 4 week supply of patches and/or lozenges dosed according to package instructions.
  Proactive telephone coaching: Patients who report continued smoking at Early (4-week) or Late (8-week) assessment of response will be randomized to receive proactive telephone coaching or not. Proactive coaching will consist of an attempt to reach the patient by telephone in order to review quit activities, provide information about locally available pharmacologic and behavioral treatment options and information sharing with patient's primary care provider. The coach is trained in core Tobacco Treatment Specialist activities.
- Late Assessment: Participants are assessed for response to brief telephone advice plus a tailored text message program at 8 weeks post-randomization. Response is based on self-reported 7-day point prevalence abstinence. Those who continue to smoke are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of of mailed NRT plus proactive telephone coaching.
  Brief telephone advice plus tailored text messages: All patients are offered brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training and a text message program tailored to readiness to quit.
  Mailed nicotine replacement therapy: Patients who report continued smoking at Early or Late assessment (depending on random assignment) will be offered a 4 week supply of patches and/or lozenges dosed according to package instructions.
  Proactive telephone coaching: Patients who report continued smoking at Early (4-week) or Late (8-week) assessment of response will be randomized to receive proactive telephone coaching or not. Proactive coaching will consist of an attempt to reach the patient by telephone in order to review quit activities, provide information about locally available pharmacologic and behavioral treatment options and information sharing with patient's primary care provider. The coach is trained in core Tobacco Treatment Specialist activities.
- Early Assessment Non-responders NRT; Early Assessment Non-responders NRT Plus Coaching; Late Assessment Non-responders NRT Plus Coaching: Individuals reporting past 7 day smoking at 4 weeks post-enrollment, randomized a second time to 4 weeks of NRT or 4 weeks of NRT plus brief telephone coaching
- Late Assessment Non-responders NRT: Individuals reporting past 7 day smoking at 8 weeks post-enrollment, randomized a second time to 4 weeks of NRT or 4 weeks of NRT plus brief telephone coaching
- Early Assessment Responders: Individuals reporting past 7 day abstinence from cigarettes at 4 weeks post-enrollment, assigned to continue text messages
- Late Assessment Responders: Individuals reporting past 7 day abstinence from cigarettes at 8 weeks post-enrollment, assigned to continue text messages
Period: Pre-assessment and Adaptation
Arm/Group | Early Assessment | Late Assessment | Early Assessment Non-responders NRT | Early Assessment Non-responders NRT Plus Coaching | Late Assessment Non-responders NRT | Late Assessment Non-responders NRT Plus Coaching | Early Assessment Responders | Late Assessment Responders
Started | 16 | 19 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 16 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post-assessment and Adaptation
Arm/Group | Early Assessment | Late Assessment | Early Assessment Non-responders NRT | Early Assessment Non-responders NRT Plus Coaching | Late Assessment Non-responders NRT | Late Assessment Non-responders NRT Plus Coaching | Early Assessment Responders | Late Assessment Responders
Started | 0 | 0 | 8 | 6 | 8 | 7 | 2 | 0
Completed | 0 | 0 | 8 | 5 | 8 | 7 | 2 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Assessment | Late Assessment | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.5) | 51.3 (14.2) | 53.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 13 | 15 | 28
  Hispanic | 0 | 1 | 1
  arican American, Non-Hispanic | 3 | 1 | 4
  Mixed, Non-Hispanic | 0 | 1 | 1
  Other, Non-Hispanic | 0 | 1 | 1
Time to first cigarette [Count of Participants; unit: Participants]
  After 60 minutes | 1 | 5 | 6
  31-60 minutes | 3 | 3 | 6
  6-30 minutes | 10 | 5 | 15
  Within 5 minutes | 2 | 6 | 8
Ready to quit in the next 30 days [Count of Participants; unit: Participants]
  No, not ready to quit in the next 30 days | 3 | 3 | 6
  Yes, ready to quit in the next 30 days | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported 7-day Abstinence From Smoking at 12 Weeks
Description: 7-day point prevalence abstinence (0, abstinent; 1, smoking), measured as "Have you smoked cigarettes, even a puff, in the past seven days?"
Time Frame: 12 weeks post-randomization
Population: Excluding n=2 withdrawn, n=3 LTFU
Measure: Count of Participants; unit: Participants
Groups:
- Early Assessment Non-responder NRT; Early Assessment Non-responder NRT Plus Coaching: Those who continue to smoke at 4 weeks are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of mailed NRT or 4 weeks of mailed NRT plus brief telephone coaching
- Early Assessment Responder: Those reporting 7 day abstinence at 4 weeks post-enrollment, assigned to continue text messages
- Late Assessment Non-responder NRT; Late Assessment Non-responder NRT Plus Coaching: Those who continue to smoke at 8 weeks are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of mailed NRT or 4 weeks of mailed NRT plus brief telephone coaching
- Late Assessment Responder: Those reporting 7 day abstinence at 8 weeks post-enrollment, assigned to continue text messages.
Arm/Group | Early Assessment Non-responder NRT | Early Assessment Non-responder NRT Plus Coaching | Early Assessment Responder | Late Assessment Non-responder NRT | Late Assessment Non-responder NRT Plus Coaching | Late Assessment Responder
Number analyzed (Participants) | 8 | 5 | 2 | 8 | 7 | 0
Participants
  0-abstinent | 0 | 1 | 1 | 4 | 1 | 0
  1-smoking | 8 | 4 | 1 | 4 | 6 | 0

2. Secondary Outcome: Number of Participants With Self-reported 7-day Abstinence From Smoking at 8 Weeks
Description: 7-day point prevalence abstinence (0, abstinent; 1, smoking)
Time Frame: 8 weeks post-randomization
Population: No participants in the late assessment group reported 7 day abstinence (all reported continued smoking) at the 8 week time point.
Measure: Count of Participants; unit: Participants
Groups:
- Early Assessment Responder: Those reporting 7 day abstinence at 4 weeks post-enrollment, assigned to continued text messages.
- Late Assessment Responder: Those reporting 7 day abstinence at 8 weeks post-enrollment, assigned to continued text messages
Arm/Group | Early Assessment Non-responder NRT | Early Assessment Non-responder NRT Plus Coaching | Early Assessment Responder | Late Assessment Non-responder NRT | Late Assessment Non-responder NRT Plus Coaching | Late Assessment Responder
Number analyzed (Participants) | 8 | 5 | 2 | 8 | 7 | 0
Participants
  0-abstinent | 0 | 1 | 2 | 0 | 0 | 0
  1-smoking | 8 | 5 | 2 | 8 | 7 | 0

3. Secondary Outcome: Exhaled Carbon Monoxide Less Than 8 Parts Per Million
Description: Exhaled carbon monoxide measured in parts per million collected at 12 weeks after enrollment
Time Frame: 12 weeks post-randomization
Population: There were no participants in the late assessment group who reported 7 day abstinence at the 8 week assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Assessment Non-responder NRT | Early Assessment Non-responder NRT Plus Coaching | Early Assessment Responder | Late Assessment Non-responder NRT | Late Assessment Non-responder NRT Plus Coaching | Late Assessment Responder
Number analyzed (Participants) | 8 | 5 | 2 | 8 | 7 | 0
Participants
  0-no biochemically verified abstinence | 8 | 4 | 1 | 5 | 6 | 0
  1-biochemically verified abstinence | 0 | 1 | 1 | 3 | 1 | 0

4. Secondary Outcome: Self-reported Number of Days Nicotine Lozenge and/or Patch Used
Description: Number of days when patch and/or lozenge was used
Time Frame: 12 weeks post-randomization
Population: Analysis compares those randomized to NRT in the second period with those randomized to NRT plus coaching in the second period, pooling early and late assessment arms together for this analysis. Excludes n=2 withdrawn, n=2 quit before second randomization, and n=2 LTFU before second randomization
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Mailed 4-week Supply of Combination NRT: Participants are assessed for response to brief telephone advice plus a tailored text message program at 4 weeks post-randomization. Response is based on self-reported 7-day point prevalence abstinence. Those who continue to smoke are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of mailed NRT plus proactive telephone coaching.
  Brief telephone advice plus tailored text messages: All patients are offered brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training and a text message program tailored to readiness to quit.
  Mailed nicotine replacement therapy: Patients who report continued smoking at Early or Late assessment (depending on random assignment) will be offered a 4 week supply of patches and/or lozenges dosed according to package instructions.
  Proactive telephone coaching: Patients who report continued smoking at Early (4-week) or Late (8-week) assessment of response will be randomized to receive proactive telephone coaching or not. Proactive coaching will consist of an attempt to reach the patient by telephone in order to review quit activities, provide information about locally available pharmacologic and behavioral treatment options and information sharing with patient's primary care provider. The coach is trained in core Tobacco Treatment Specialist activities.
- Mailed 4-week Supply of Combination NRT Plus Proactive Telephone Coaching: Participants are assessed for response to brief telephone advice plus a tailored text message program at 8 weeks post-randomization. Response is based on self-reported 7-day point prevalence abstinence. Those who continue to smoke are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of of mailed NRT plus proactive telephone coaching.
  Brief telephone advice plus tailored text messages: All patients are offered brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training and a text message program tailored to readiness to quit.
  Mailed nicotine replacement therapy: Patients who report continued smoking at Early or Late assessment (depending on random assignment) will be offered a 4 week supply of patches and/or lozenges dosed according to package instructions.
  Proactive telephone coaching: Patients who report continued smoking at Early (4-week) or Late (8-week) assessment of response will be randomized to receive proactive telephone coaching or not. Proactive coaching will consist of an attempt to reach the patient by telephone in order to review quit activities, provide information about locally available pharmacologic and behavioral treatment options and information sharing with patient's primary care provider. The coach is trained in core Tobacco Treatment Specialist activities.
Arm/Group | Mailed 4-week Supply of Combination NRT | Mailed 4-week Supply of Combination NRT Plus Proactive Telephone Coaching
Number analyzed (Participants) | 16 | 13
Days | 5.8 (2.4) | 7.0 (0.0)

5. Secondary Outcome: Self-reported Change in Average Number of Cigarettes Smoked Per Day
Description: Self-reported change in average cigarettes smoked per day
Time Frame: 12 weeks post-randomization
Population: No participants randomized to late assessment reported 7 day abstinence at 8 weeks post-enrollment.
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Early Assessment Non-responder NRT | Early Assessment Non-responder NRT Plus Coaching | Early Assessment Responder | Late Assessment Non-responder NRT | Late Assessment Non-responder NRT Plus Coaching | Late Assessment Responder
Number analyzed (Participants) | 8 | 5 | 2 | 8 | 7 | 0
Cigarettes per day | -7.0 (7.3) | -7.2 (7.7) | -13.0 (9.9) | -12.5 (9.3) | -4.7 (7.3) |

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Early Assessment Non-responder NRT; Early Assessment Non-responder NRT Plus Coaching: Participants are assessed for response to brief telephone advice plus a tailored text message program at 4 weeks post-enrollment. Response is based on self-reported 7-day point prevalence abstinence. Those who continue to smoke are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of mailed NRT plus proactive telephone coaching.
  Brief telephone advice plus tailored text messages: All patients are offered brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training and a text message program tailored to readiness to quit.
  Mailed nicotine replacement therapy: Patients who report continued smoking at Early or Late assessment (depending on random assignment) will be offered a 4 week supply of patches and/or lozenges dosed according to package instructions.
  Proactive telephone coaching: Patients who report continued smoking at Early (4-week) or Late (8-week) assessment of response will be randomized to receive proactive telephone coaching or not. Proactive coaching will consist of an attempt to reach the patient by telephone in order to review quit activities, provide information about locally available pharmacologic and behavioral treatment options and information sharing with patient's primary care provider. The coach is trained in core Tobacco Treatment Specialist activities.
- Early Assessment Responder: Reported 7 day abstinence at 4 weeks post-enrollment, assigned to continue text messages.
- Late Assessment Non-responder NRT; Late Assessment Non-responder NRT Plus Coaching: Participants are assessed for response to brief telephone advice plus a tailored text message program at 8 weeks post-enrollment. Response is based on self-reported 7-day point prevalence abstinence. Those who continue to smoke are randomized to the offer of 4 week supply of mailed nicotine patches and/or lozenges (NRT) or 4 week supply of of mailed NRT plus proactive telephone coaching.
  Brief telephone advice plus tailored text messages: All patients are offered brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training and a text message program tailored to readiness to quit.
  Mailed nicotine replacement therapy: Patients who report continued smoking at Early or Late assessment (depending on random assignment) will be offered a 4 week supply of patches and/or lozenges dosed according to package instructions.
  Proactive telephone coaching: Patients who report continued smoking at Early (4-week) or Late (8-week) assessment of response will be randomized to receive proactive telephone coaching or not. Proactive coaching will consist of an attempt to reach the patient by telephone in order to review quit activities, provide information about locally available pharmacologic and behavioral treatment options and information sharing with patient's primary care provider. The coach is trained in core Tobacco Treatment Specialist activities.
Arm/Group | Early Assessment Non-responder NRT | Early Assessment Non-responder NRT Plus Coaching | Early Assessment Responder | Late Assessment Non-responder NRT | Late Assessment Non-responder NRT Plus Coaching
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/2 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/2 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 2/5 | 0/2 | 1/8 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Assessment Non-responder NRT (N=8) | Early Assessment Non-responder NRT Plus Coaching (N=5) | Early Assessment Responder (N=2) | Late Assessment Non-responder NRT (N=8) | Late Assessment Non-responder NRT Plus Coaching (N=7)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiccup (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild anxiety

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT04020718/Prot_SAP_000.pdf